CLINICAL TRIAL: NCT06328465
Title: fREEDOM: REsonance for Early Detection Of Breast Cancer Metastases
Acronym: fREEDOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UID 1743; IEO 1108 (Other: Comitato Etico degli IRCCS Istituto Europeo di Oncologia e Centro Cardiologico Monzino)
Record Dates: First submitted 2024-03-13; First posted 2024-03-25 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Invasive Breast Cancer; HER2-positive Breast Cancer; Triple Negative Breast Cancer
Keywords: Invasive Breast Cancer; HER2-positive Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DWB-MRI (Experimental): Surveillance with diffusion whole body MRI
  Interventions: Diagnostic Test: Diffusion whole body MRI

INTERVENTIONS:
Diagnostic Test: Diffusion whole body MRI — Diffusion whole body MRI protocol, consisting of sagittal T1-weighted and T2-weighted sequences on the whole spine, axial T1 weighted, T2-weighted and diffusion-weighted images from head to mid-thigh, performed on a 1.5 T scanner.

SUMMARY:
The aim of this study is to understand whether DWB-MRI (Diffusion Whole Body-Magnetic Resonance Imaging) is useful for early detection of locoregional or distant recurrence and whether early diagnosis influences the prognosis in high-risk populations thanks to the possibility of being able to use a more effective treatment. The primary objective is to evaluate 5-year overall survival (OS) in patients with Human Epidermal Growth Factor Receptor 2 positive (HER2+) or high-risk Triple Negative (TN) undergoing surveillance with DWB-MRI.

DETAILED DESCRIPTION:
Breast cancer is the second most common cancer in the world and the most common cancer among women. In these patients, it is not the primary tumor, but its distant metastases that are the main cause of death. Follow-up may vary depending on the hospital or doctor, but the data available in the literature do not show an advantage in terms of survival or quality of life in patients subjected to intensive follow-up. However, the information that physicians have comes from past studies limited by the presence of bias regarding patient characteristics, therapies, follow-up intervals and tests used. In light of the better understanding of biology, breast cancer is no longer considered a single disease, but it is classified into at least four different molecular subtypes, based on the immunohistochemical classification: Luminal A-like, Luminal B-like, HER2 positive and Triple Negative. Nowadays it is known that not only the stage of diagnosis, but also the biology of the disease influences the risk of recurrence and death. Furthermore, a growing number of trials show that different biological subtypes differ in terms of time to relapse and disease pattern of metastatic spread (in particular, site of first relapse). These observations lead to the hypothesis that different types and different frequencies of follow-up strategies should vary depending on the biology of breast cancer. Furthermore, with improved management and the availability of new effective treatments, patients with oligometastatic disease treated with an aggressive multidisciplinary approach may be amenable to curative treatment. Based on this hypothesis, an early diagnosis of metastatic disease could lead to the identification of patients with low disease burden who can still be treated with curative intent. DWB-MRI is emerging as a promising tool for the detection and therapy monitoring of metastases in different tumor types and could be an important tool for the early detection of breast cancer metastases.

ELIGIBILITY:
Inclusion Criteria:

* Pre or post-menopausal patient with histologically confirmed invasive breast cancer stage II - III HER2 + or TN operated breast carcinoma or patients underwent neoadjuvant treatment (included cT4d) with residual disease at definitive surgery
* No evidence of distant metastases at baseline perioperative radiological staging (DWB-MRI, total body Computed Tomography (CT) or Positron Emission Tomography (PET/CT) must be performed +/- 1 month from surgery)
* No relevant comorbidities
* Eastern Cooperative Oncology Group (ECOG) performance status 0
* Geographically accessible for follow up
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Absolute contraindications that exclude the execution of the MRI investigation, regardless of the clinical indication
* Relative contraindications that include situations in which the innocuousness of the examination is not documented with certainty that therefore do not recommend the execution, except for serious indications related to the patient's clinical need
* Older age (>75 years)
* Previous or concomitant other malignancy except basal or squamous cell carcinoma of the skin or adequately treated in situ carcinoma of the cervix
* Uncontrolled intercurrent illness including symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 years
  Number of alive patients at 5 years (considering deaths from any cause)

SECONDARY OUTCOMES:
Overall survival of patients underwent local treatment | 5 years
  Number of patients undergoing local treatment (surgery or other localized technique) who are alive at 5 years (considering deaths from any cause)
Breast cancer specific survival | 5 years
  Number of alive patients at 5 years (considering only deaths related to breast cancer)
Safety of local treatment | 48 months
  Number of serious adverse event related to local treatment received
Anxiety assessment | 48 months
  Collection of Hamilton Anxiety Rating Scale questionnaire (minimum value: 0, maximum value: 4 - higher scores mean a worse outcome)
Health state assessment | 48 months
  Collection of 12-Item Short Form Survey (SF-12) questionnaire (minimum value: 0, maximum value: 6 - higher scores mean a better outcome)
Ability to Cope With Trauma assessment | 48 months
  Collection of Perceived Ability to Cope With Trauma (PACT) questionnaire (minimum value: 0, maximum value: 7 - higher scores mean a better outcome)
Personality assessment | 48 months
  Collection of Big Five Personality Inventory (BFI-10) questionnaire (minimum value: 0, maximum value: 5 - higher scores mean a greater agreement with the statement)
Acceptability and perception of DWB-MRI | 48 months
  Collection of Acceptance Questionnaire (minimum value: 0, maximum value: 5 - higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Iorfida, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy